CLINICAL TRIAL: NCT00474799
Title: An Open Label, Randomized, Single Center, Repeat Dose Study to Assess the Safety, Tolerability and Pharmacokinetic Profile of MNS075 (Intranasal Morphine) in Opioid naïve, Healthy Adult Volunteers
Brief Title: Study to Assess the Safety, Tolerability and Pharmacokinetic Profile of MNS075 (Intranasal Morphine)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Javelin Pharmaceuticals (Industry)
Responsible Party: Javelin Pharmaceuticals, Javelin Pharmaceuticals
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: MOR-PK-006
Record Dates: First submitted 2007-05-15; First posted 2007-05-17 (Estimated); Last update posted 2008-01-14 (Estimated); Status verified 2008-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): MNS075 7.5mg q1h
  Interventions: Drug: MNS075
- B (Experimental): MNS075 15mg q3h
  Interventions: Drug: MNS075

INTERVENTIONS:
Drug: MNS075 — MNS075 7.5mg q1h MNS075 15mg q3h

SUMMARY:
The purpose of this study is to characterize the repeat dosing plasma profile, extent of accumulation and repeat dose pharmacokinetics of morphine, morphine-3-glucuronide, and morphine-6-glucuronide during administration of MNS075 in two different, clinically-relevant dosing schedules.

DETAILED DESCRIPTION:
This study is an open label, randomized, two-treatment, two-period, two-sequence, single-center, crossover study comparing the pharmacokinetics, safety and tolerability of MNS075 (intranasal morphine) at doses of 7.5 mg self-administered q1h for 7 hours (8 doses) and 15 mg self-administered q3h for 9 hours (4 doses).

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers 18 years of age or older

Exclusion Criteria:

* History of alcohol, drug addiction, or substance abuse.
* Known to or suspected to be currently abusing alcohol or drugs.
* Allergy or hypersensitivity to shellfish or opioids.
* History of seizures.
* Clinically significant structural or functional abnormalities of the nose and upper airway, obstruction of the nasal passages, or mucosal lesions of the nostrils.
* Smoked or used tobacco or nicotine products in the past six months or expects to during the study.
* Positive for hepatitis B or hepatitis C or HIV antibodies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-01; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
To characterize the repeat dosing plasma profile, extent of accumulation and repeat dose pharmacokinetics of morphine, morphine-3-glucuronide, and morphine-6-glucuronide during administration of MNS075. | Multiple

CONTACTS AND LOCATIONS:
Overall Officials: Javelin Pharmaceuticals, Study Director — Javelin Pharmaceuticals
Locations (1):
- CEDRA Corporation, Austin, Texas, United States